CLINICAL TRIAL: NCT00444171
Title: Randomized Controlled Trial to Evaluate Blood Glucose Control by the Model Predictive Control Algorithm With Variable Sampling Rate (eMPC) vs. Routine Glucose Management Protocol in Peri- and Postoperative Period in Cardiac Surgery Patients
Brief Title: Glucose Control by eMPC Algorithm in Peri- and Postoperative Period in Cardiac Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: eMPC_CUP1
Record Dates: First submitted 2007-03-05; First posted 2007-03-07 (Estimated); Last update posted 2007-03-07 (Estimated); Status verified 2007-03

CONDITIONS: Cardiac Surgery Patients; Blood Glucose
Keywords: critically ill; insulin resistance; intensive insulin therapy; computer algorithm
MeSH Terms: conditions — Critical Illness; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: insulin infusion rate controled by computer algorithm
Procedure: insulin infusion rate guided by in-house glucose management protocol

SUMMARY:
Randomized controlled trial to compare blood glucose control by the model predictive control algorithm with variable sampling rate (eMPC) with routine glucose management protocol (RMP) in peri- and postoperative period in cardiac surgery patients.

DETAILED DESCRIPTION:
Context. Increased blood glucose levels frequently occur in critically ill patients and its normalization by intensive insulin treatment markedly improves clinical outcome.

Objective and Design: Randomized controlled trial to compare blood glucose control by the model predictive control algorithm with variable sampling rate (eMPC) with routine glucose management protocol (RMP) in peri- and postoperative period in cardiac surgery patients.

Setting: Department of Cardiac Surgery, University Hospital. Patients. 60 cardiac surgery patients. Interventions. Elective cardiac surgery and treatment with continuous insulin infusion to maintain euglycemia (target range 4.4 - 6.1 mmol/l). 30 patients were randomized for eMPC and 30 for RMP treatment. Blood glucose was measured in 1-4 hour intervals depending on request of each algorithm during surgery and post-operation period for 24 hours.

Main Outcome Measures. Mean blood glucose, percentage of time in target range. Results. Mean blood glucose was 6.15 ± 1.11 mmol/l in eMPC vs. 7.21 ± 1.08 mmol/l in RMP group (p<0.05); percentage of time in target range was 60.4 ± 22.8% for eMPC vs. 27.5 ± 16.2% for RMP group (p<0.05). No severe hypoglycemia (blood glucose bellow 2.9 mmol/l) was observed during the study. Average insulin infusion rate was 4.67 ± 3.34 in eMPC vs. 2.57 ± 1.66 IU/h in RMP (p<0.05), average sampling interval was 1.46 ± 0.31 vs. 2.10 ± 0.22 hours (p<0.05).

Conclusions. eMPC algorithm was more effective and comparably safe as compared to RMP in maintaining euglycemia in cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Elective cardiac surgery

Exclusion Criteria:

* Allergy against insulin
* Mental incapacity
* Language barrier

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2006-09; Study Completion 2007-02

PRIMARY OUTCOMES:
Mean blood glucose
percentage of time in target range

SECONDARY OUTCOMES:
Number of hypoglycaemic episodes

CONTACTS AND LOCATIONS:
Overall Officials: Stepan Svacina, MD, DSc, Principal Investigator — Charles University Prague
Locations (1):
- General University Hospital, Prague, Czechia